CLINICAL TRIAL: NCT01314716
Title: A Phase 3, Double-Blind, Multicenter, Randomized, Placebo-Controlled Trial Evaluating Repeated Courses of Aztreonam for Inhalation Solution/Aztreonam 75 mg Powder and Solvent for Nebuliser Solution in Subjects With Non-CF Bronchiectasis and Gram-Negative Endobronchial Infection (AIR-BX2)
Brief Title: Safety and Effectiveness of AZLI (an Inhaled Antibiotic) in Adults With Non-Cystic Fibrosis Bronchiectasis
Acronym: AIR-BX2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-219-0104
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZLI-AZLI (Experimental): Participants were randomized to receive blinded AZLI for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI for 28 days plus 56 days of treatment-free follow-up.
  Interventions: Drug: AZLI
- Placebo-AZLI (Placebo Comparator): Participants were randomized to receive blinded placebo to match AZLI for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI for 28 days plus 56 days of treatment-free follow-up.
  Interventions: Drug: AZLI; Drug: Placebo

INTERVENTIONS:
Drug: AZLI — AZLI 75 mg reconstituted with diluent and administered via nebulizer three times daily
Drug: Placebo — Placebo to match AZLI administered via nebulizer three times daily
  Arms: Placebo-AZLI

SUMMARY:
The AIR-BX2 study enrolled people with non-cystic fibrosis (non-CF) bronchiectasis and gram-negative airway infection. Participants received two 28-day courses of either Aztreonam for Inhalation Solution (AZLI) or placebo taken 3 times a day. Each course was followed by a 28-day off-drug period. Following the two blinded courses, all participants received a 28-day course of open-label AZLI then were followed for an additional 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female 18 years or older with non-CF bronchiectasis
* Chronic sputum production on most days
* Positive sputum culture for gram-negative organisms
* Must have met lung function requirements

Exclusion Criteria:

* History of CF
* Hospitalized within 14 days prior to joining the study
* Previous exposure to AZLI
* Pregnant, breastfeeding, or unwilling to follow contraceptive measures for the study
* Must have met liver and kidney function requirements
* Continuous oxygen use of greater than 2 liters per minute (supplemental oxygen with activity and at night was allowed)
* Treatment for nontuberculous mycobacteria infection or active mycobacterium tuberculosis infection within 1 year of enrollment
* Other serious medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne O'Donnell, MD, Principal Investigator — Georgetown University Hospital
Locations (85):
- United States (33):
  - Florence Research Associates, Florence, Alabama
  - Clinical Trials Connection, Flagstaff, Arizona
  - Phoenix Medical Group, Peoria, Arizona
  - Pulmonary Associates, Phoenix, Arizona
  - AZ Pulmonary Specialists, LTD, Scottsdale, Arizona
  - Pulmonary Consultants & Primary Care Physicians Medical Group, Inc., Orange, California
  - UC San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Sarasota Memorial Hospital - Clinical Research Center, Sarasota, Florida
  - Pasadena Center for Medical Research, St. Petersburg, Florida
  - Tampa General Hospital - New Lung Associates, Tampa, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Southeastern Lung Care PC, Decatur, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loess Hills Clinical Research, Council Bluffs, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Pulmonary & Critical Care Associates of Baltimore, Rosedale, Maryland
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Pulmonary & Allergy Associates, P.A., Summit, New Jersey
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Columbia University, NY Presbyterian Hospital, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - The Oregon Clinic P.C./ Pulmonary Division, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Pulmonary Consultants, PLLC, Tacoma, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Australia (9):
  - Concord Hospital, Concord, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Royal Perth Hospital, Perth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Repatriation General Hospital, Daw Park, South Australia
  - Burnside War Memorial Hospital Pharmacy, Toorak Gardens, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (3):
  - CUB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - KUL UZ Gasthuisberg, Leuven
- Canada (3):
  - Kelowna Respiratory Research and Allergy Clinic, Kelowna, British Columbia
  - The Lung Centre at Vancouver General Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
- France (6):
  - CHICAS - Centre Hospitalier Intercommunal des Alpes du sud, site de GAP, Gap, PACA
  - Service Activite Ambulatoire Pole Cardiovasculaire Hopital Nord, Marseille
  - CHU de Montpellier-Hopital Arnaud de Villeneuve, Montpellier
  - Hôpital Pasteur, CHU de Nice, Nice
  - Hopital Haut-Leveque, Pessac
  - CHU Toulouse - Hôpital Larrey, Toulouse
- Germany (10):
  - Charite Campus Virchow-Klinikum, Berlin
  - Research Center for Medical Studies (RCMS), Berlin-Charlottenburg (Westend)
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - University Hospital Giessen, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena Clinic for Internal Medicine II, Jena
  - Univ.-Klinikum Leipzig, Innere Med., Leipzig
  - POIS Leipzig GbR, Leipzig
  - Klinikum Innenstadt der LMU Munchen, Munich
- Italy (6):
  - S.Anna Hospital, University of Ferrara, Ferrara
  - UO Broncopneumologia IRCCS Fondazione Cà Granda Milano, Milan
  - University of Modena and Reggio Emilia, Modena
  - Azienda Universitaria Federico II, Naples
  - Università di Pisa - Ospedale Cisanello, Pisa
  - Ospendale Civile Maggiore Centro Regionale Fibrosi Cistica, Verona
- Netherlands (2):
  - Medisch Centrum Alkmaar, Alkmaar
  - Erasmus MC, Rotterdam
- Spain (6):
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Universitario La Paz, Madrid
  - Hospital La Fe, Valencia
- United Kingdom (7):
  - Papworth Hospital NHS Trust, Cambridgeshire
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, NHS Foundation Trust, Exeter
  - Sir William Leech Centre for Lung Research, Freeman Hospital, Newcastle upon Tyne
  - GBS RE Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Torbay District General Hospital, Torquay, Devon
  - Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Barker AF, O'Donnell AE, Flume P, Thompson PJ, Ruzi JD, de Gracia J, Boersma WG, De Soyza A, Shao L, Zhang J, Haas L, Lewis SA, Leitzinger S, Montgomery AB, McKevitt MT, Gossage D, Quittner AL, O'Riordan TG. Aztreonam for inhalation solution in patients with non-cystic fibrosis bronchiectasis (AIR-BX1 and AIR-BX2): two randomised double-blind, placebo-controlled phase 3 trials. Lancet Respir Med. 2014 Sep;2(9):738-49. doi: 10.1016/S2213-2600(14)70165-1. Epub 2014 Aug 18. PMID 25154045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 90 study sites in the North America, Europe, and Australia. The first participant was screened on 25 April 2011. The last participant observation was on 01 July 2013.
Pre-assignment Details: 404 participants were screened, 274 were randomized and comprise the Intent-to-Treat (ITT) Analysis Set. 272 randomized participants received at least one dose of study drug and comprise the Safety Analysis Set.
Groups:
- AZLI-AZLI: Participants were randomized to receive blinded Aztreonam for Inhalation Solution (AZLI) 75 mg three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 84 days.
- Placebo-AZLI: Participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 84 days.
Period: Double-Blind Phase
Arm/Group | AZLI-AZLI | Placebo-AZLI
Started | 136 | 138
Randomized and Treated | 135 | 137
Completed | 119 | 123
Not Completed | 17 | 15
Not completed — Randomized but not treated | 1 | 1
Not completed — Adverse Event | 10 | 4
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor request | 1 | 2
Not completed — Physician Decision | 0 | 1
Period: Open-Label Phase
Arm/Group | AZLI-AZLI | Placebo-AZLI
Started | 112 (7 participants in this group did not continue from the randomized to the open-label phase.) | 110 (13 participants in this group did not continue from the randomized to the open-label phase.)
Completed | 102 | 98
Not Completed | 10 | 12
Not completed — Adverse Event | 4 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 5 | 4

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- AZLI-AZLI: Participants were randomized to receive blinded AZLI 75 mg three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Placebo-AZLI: Participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each cycle followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Total: Total of all reporting groups
Arm/Group | AZLI-AZLI | Placebo-AZLI | Total
Number analyzed (Participants) | 136 | 138 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (14.22) | 62.7 (13.33) | 63.0 (13.75)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 66 | 119
  >=65 years | 83 | 72 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 101 | 190
  Male | 47 | 37 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 122 | 112 | 234
  Unknown or Not Reported | 9 | 19 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 119 | 128 | 247
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Black or African Heritage | 2 | 4 | 6
  Other | 2 | 1 | 3
  Not permitted | 11 | 4 | 15
Region of Enrollment [Number; unit: participants]
  France | 11 | 3 | 14
  United States | 58 | 52 | 110
  Canada | 0 | 2 | 2
  Spain | 22 | 17 | 39
  Belgium | 5 | 6 | 11
  Australia | 3 | 2 | 5
  Netherlands | 5 | 12 | 17
  Germany | 16 | 21 | 37
  United Kingdom | 11 | 11 | 22
  Italy | 5 | 12 | 17
QOL-B Respiratory Symptom Score [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Questionnaire-Bronchiectasis (QOL-B) overall score was scaled from 0-100 with higher scores representing better quality of life.
  units on a scale | 56.2 (17.98) | 57.4 (18.07) | 56.8 (18.00)

OUTCOME MEASURES:

1. Primary Outcome: Change in QOL-B Respiratory Symptoms Score at Day 28
Description: The mean (SD) change in the Respiratory Symptoms score on the Quality of Life Questionnaire-Bronchiectasis (QOL-B) was measured from baseline to the end of Course 1 (Day 28). The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Time Frame: Baseline to Day 28
Population: Participants in the ITT Analysis Set with scores at both baseline and Day 28 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 128 | 132
units on a scale | 8.2 (17.13) | 3.2 (14.67)
Statistical Analysis 1: Comparison: AZLI-AZLI vs Placebo-AZLI; Test type: Superiority or Other; p = 0.011, MMRM — P-value was based on T-test from mixed-effect model repeated measures (MMRM); Differences in least squares mean = 4.6, 95% CI 2-sided [1.1 to 8.2]

2. Secondary Outcome: Change in QOL-B Respiratory Symptoms Score at Day 84
Description: The mean (SD) change in the Respiratory Symptoms score on the QOL-B was measured from baseline to the end of Course 2 (Day 84). The QOL-B respiratory symptoms score was transformed onto a scale of 0-100, with higher scores representing a better quality of life.
Time Frame: Baseline to Day 84
Population: Participants in the ITT Analysis Set with scores at both baseline and Day 84 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 123 | 125
units on a scale | 5.6 (16.44) | 3.9 (17.73)
Statistical Analysis 1: Comparison: AZLI-AZLI vs Placebo-AZLI; Test type: Superiority or Other; p = 0.56, MMRM — P-value was based on T-test from mixed-effect model repeated measures (MMRM); Difference in least squares mean = 1.1, 95% CI 2-sided [-2.7 to 5.0]

3. Secondary Outcome: Time to Protocol-Defined Exacerbation (PDE)
Description: Protocol-defined exacerbation was defined as an acute worsening of respiratory disease that triggered the initiation of a non-study antibiotic meeting at least 3 major criteria, or 2 major and at least 2 minor criteria.
  * Major Criteria: increased sputum production; increased discoloration of sputum; increased dyspnea; increased cough
  * Minor Criteria: fever (> 38º C) measured during clinic visit; increased malaise or fatigue; forced expiratory volume in 1 second (FEV1) (L) or forced vital capacity (FVC) decreased > 10% from baseline; new or increased hemoptysis
Time Frame: Baseline to Day 112
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI-AZLI | Placebo-AZLI
Number analyzed (Participants) | 136 | 138
days | NA [NA to NA] — At least 50% of participants must have had a PDE in order to compute the median days to PDE. Fewer than 50% of participants in this group had a PDE, so median days to PDE could not be computed. | NA [NA to NA] — At least 50% of participants must have had a PDE in order to compute the median days to PDE. Fewer than 50% of participants in this group had a PDE, so median days to PDE could not be computed.

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug
Groups:
- AZLI-AZLI (Double-Blind): Adverse events for this reporting group were reported from baseline to Day 112 while participants were receiving double-blind AZLI; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- Placebo-AZLI (Double-Blind): Adverse events for this reporting group were reported from baseline to Day 112 while participants were receiving double-blind placebo; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
- AZLI-AZLI (Open-Label); Placebo-AZLI (Open-Label): Adverse events for this reporting group were reported from Day 112 to Day 196 plus 30 days while participants were receiving open-label AZLI; participants were randomized to receive blinded placebo to match AZLI three times daily via investigational nebulizer for 2 cycles of 28 days on treatment with each followed by 28 days off treatment, followed by open-label AZLI 75 mg three times daily for 28 days plus 56 days of treatment-free follow-up.
Arm/Group | AZLI-AZLI (Double-Blind) | Placebo-AZLI (Double-Blind) | AZLI-AZLI (Open-Label) | Placebo-AZLI (Open-Label)
Serious Adverse Events (participants affected / at risk) | 18/135 | 16/137 | 8/112 | 9/110
Other Adverse Events (participants affected / at risk) | 112/135 | 101/137 | 54/112 | 58/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI-AZLI (Double-Blind) (N=135) | Placebo-AZLI (Double-Blind) (N=137) | AZLI-AZLI (Open-Label) (N=112) | Placebo-AZLI (Open-Label) (N=110)
Infective exacerbation of bronchiectasis (Infections and infestations) | 4 | 2 | 0 | 3
Pneumonia (Infections and infestations) | 3 | 2 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI-AZLI (Double-Blind) (N=135) | Placebo-AZLI (Double-Blind) (N=137) | AZLI-AZLI (Open-Label) (N=112) | Placebo-AZLI (Open-Label) (N=110)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 65 | 27 | 38
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 59 | 50 | 19 | 23
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 48 | 38 | 21 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 47 | 26 | 28
Wheezing (Respiratory, thoracic and mediastinal disorders) | 18 | 13 | 11 | 7
Fatigue (General disorders) | 25 | 25 | 14 | 16
Malaise (General disorders) | 14 | 19 | 4 | 6
Pyrexia (General disorders) | 30 | 21 | 12 | 16
Non-cardiac chest pain (General disorders) | 9 | 13 | 5 | 10
Headache (Nervous system disorders) | 17 | 14 | 7 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0 | 0
Chills (General disorders) | 10 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 7 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 7 | 0 | 0
Pain (General disorders) | 0 | 0 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years